CLINICAL TRIAL: NCT01001000
Title: Colour Coded Duplex Ultrasound of Native Arterio-venous Fistula for Haemodialysis With Venous Pressure Measurement Using Controlled Compression Ultrasound as a Predictor for Shunt Maturation in the Early Postoperative Phase
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Christoph Thalhammer, MD, USZ
Other Study IDs: CT-01-2009-USZ
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Ultrasound (Pressure measurement) — cut-off value for non maturationg fistulas

SUMMARY:
Prospective observational ultrasound study of native arterio-venous fistula for haemodialysis with venous pressure measurement using controlled compression ultrasound.

ELIGIBILITY:
Inclusion criteria:

* Patients after creation of a native arterio-venous fistula at the cephalic vein for hemodialysis access;
* Informed consent.

Exclusion criteria:

* Former creation of a native arterio-venous fistula at the same arm;
* Known upper extremity occlusive arterial disease;
* Situation when ultrasound examination is not suitable: extreme swelling of the arm, post-operative pain, hematoma, local infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after creation of a native arterio-venous fistula at the cephalic vein for hemodialysis access
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-10; Study Completion 2010-10

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland